CLINICAL TRIAL: NCT05002842
Title: Implementation of Mind-Body Practices in an Online Community of Caring (CaringBridge)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 1703S09842
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Cancer; Stress
Keywords: Cancer; Gratitude; Social Support; Online; Perceived Stress; CaringBridge; Social Connectedness; Social Assurance
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): Those in the immediate intervention arm will begin the LovingKindess Meditation practice upon enrollment.
  Interventions: Behavioral: LovingKindess Meditation
- Delayed Intervention (Experimental): Those in the deferred intervention arm will commence the LovingKindness Meditation practice intervention approximately 3 weeks (post 3 -week survey) after enrollment and participate three weeks thereafter.
  Interventions: Behavioral: LovingKindess Meditation

INTERVENTIONS:
Behavioral: LovingKindess Meditation — Participants will have access to a recording of a script to guide them through meditation

SUMMARY:
CaringBridge (CB) is an online health community for people undergoing challenging health journeys. This platform provides an opportunity for individuals and their caregivers to rally support for a loved-one during a health journey. CaringBridge offers the opportunity for expressive writing through journal entries, wellbeing resources, participant health journey stories, and practical scheduling and communication tools to support community, healing, and wellbeing. Loving Kindness Meditation (LKM) is a systemized mind-body approach developed to increase loving acceptance and has been shown to increase resilience in the face of adversity. The aim of this study is to better understand how mind-body practices, like LKM, impact adult CB users

ELIGIBILITY:
Inclusion Criteria:

* English literacy
* CaringBridge user with an active email address
* Visitor/Caregiver/Patient on a Cancer Journey (for Phase 2 only)

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 979 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress: The Perceived Stress Scale | 3 weeks
  The Perceived Stress Scale is a 10-item scale for measuring one's perception of stress. All 10 items are assessed by asking how often a respondent felt a certain way on a 5-point Likert measure (0 = Never; 4 = Very Often), with a minimum score of 0 and a maximum score of 40. Higher total scores indicate greater perceived stress.
  This will be assessed at baseline and week three, in addition to week six for the deferred arm.

SECONDARY OUTCOMES:
Change in Self-Compassion: The Self-Compassion Scale | 3 weeks
  The Self-Compassion Scale (SCS) is a 12-item, shortened version of the original longer 26-item self-compassion scale (range 12-60). The 12-item SCS contains the same higher-order factor structure as the 26-item scale with a general Higher-Order Self-Compassion factor and six second-order factors of Self-Kindness, Self-Judgement, Common Humanity, Isolation, Mindfulness, and Over-Identification. All 12 items are assessed by asking how often a respondent felt a certain way on a 5-point Likert measure (1 =Almost never; 5 =Almost always). Higher SCS scores are associated with psychological well-being and suggest self-compassion might be an important protective factor, fostering emotional resilience.
  This will be assessed at baseline and week three, in addition to week six for the deferred arm.
Change in Compassionate Love: The Compassionate Love for Humanity Scale | 3 weeks
  The Compassionate Love Scale (CLS) is a 21-item measure of the stranger-humanity version of the original CLS designed to measure compassionate love for humanity (range 38-147). Higher CLS scores indicate greater compassionate love for humanity.
  This will be assessed at baseline and week three, in addition to week six for the deferred arm.
Change in Social Support: The Social Connectedness Scale | 3 weeks
  Social connectedness is assessed with 8 items on a 6-point Likert scale (1 = strongly agree through 6 = strongly disagree), with a total range of 8-48. Social connectedness is reverse coded such that high scores indicate higher social connection.
  This will be assessed at baseline and week three, in addition to week six for the deferred arm.
Change in Social Support: The Social Assurance Scale | 3 weeks
  Social assurance is assessed with 8 items on a 6-point Likert scale (1 = strongly agree through 6 = strongly disagree), with a total range of 8-48. Social Assurance is reverse coded such that high scores indicate higher social assurance. This will be assessed at baseline and week three, in addition to week six for the deferred arm.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jo Kreitzer, PhD, RN, FAAN, Principal Investigator — University of Minnesota Earl E. Bakken Center for Spirituality & Healing
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Telke S, Leininger B, Hanson L, Kreitzer MJ. A Randomized Trial of 21 Days of Loving Kindness Meditation for Stress Reduction and Emotional Well-being Within an Online Health Community for Patients, Family, and Friends Experiencing a Cancer Health Journey. J Integr Complement Med. 2022 Feb;28(2):158-167. doi: 10.1089/jicm.2020.0512. Epub 2022 Jan 11. PMID 35167360